CLINICAL TRIAL: NCT02045017
Title: A Phase 2 Multicenter, Open-label Study to Determine the Efficacy and Safety of Pomalidomide (CC-4047) in Combination With Low-Dose Dexamethasone in Subjects With Relapsed or Refractory Multiple Myeloma and Moderate or Severe Renal Impairment Including Subjects Undergoing Hemodialysis
Brief Title: Efficacy and Safety of Pomalidomide and Dexamethasone in RRMM Patients With Renal Insufficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-4047-MM-013; 2013-001903-36 (EudraCT Number)
Record Dates: First submitted 2013-12-16; First posted 2014-01-24 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed Multiple Myeloma; Refactory Multiple Myeloma; Renal Insufficiency; Pomalidomide; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma; Renal Insufficiency | interventions — pomalidomide; Dexamethasone; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pomalidomide and low dose Dexamethasone (Experimental): Pomalidomide 4mg, and low dose Dexamethasone, starting at 40mgs(≤ 75 years old) or 20 mg/day (> 75 years old)
  Interventions: Drug: Pomalidomide and Dexamethasone

INTERVENTIONS:
Drug: Pomalidomide and Dexamethasone
  Other Names: Tablet

SUMMARY:
The primary purpose of the study is to determine the safety and efficacy and to generate PK and biomarker data for the combination of Pomalidomide and low-dose Dexamethasone in patients with relapsed or refractory multiple myeloma, with moderate or severe renal impairment.

DETAILED DESCRIPTION:
The study will consist of a Screening phase within 28 days prior to cycle 1 day 1. Subjects once enrolled will enter the Treatment phase, in which patients will be treated until progression, or study discontinuation due to other reasons. Subjects will enter the long term Follow-up phase of the study where data will be collected every 3 months for up to 5 years on Secondary primary malignancies, survival, subsequent anti myeloma treatments and date of progression. Subjects will be recruited into one of 3 cohorts depending on the severity of their renal impairment.

ELIGIBILITY:
Inclusion Criteria:

- Subjects must satisfy the following criteria to be enrolled in the study.

1. Subjects must have documented diagnosis of multiple myeloma and have measurable disease (serum M-protein ≥ 0.5 g/dL or urine M-protein ≥ 200 mg/24 hours).

5. Subjects must have had at least 1 prior antimyeloma regimen including lenalidomide and documented progression as per the International Myeloma Working Group uniform response criteria (Durie, 2006) during or after the last antimyeloma regimen. Induction therapy followed by Autologous Stem Cell Transplant and consolidation/ maintenance will be considered as one regimen.

6. Subjects must have an impaired renal function with an estimated Glomerular Filtrate Rate of < 45 mL/min/1.73 m2 according to the modification of diet in renal disease equation.

1. Impaired renal function must be due to multiple myeloma which needs to be confirmed by kidney biopsy.
2. Subjects may have acute myeloma related renal failure or chronic myeloma related renal failure; they may also have been treated with dialysis before, including dialysis with high cut off membranes.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment

1. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Renal insufficiency due to other reasons than multiple myeloma or due to hypocalcaemia only.
4. Prior history of malignancies, other than MM, unless the subject has been free of the disease for ≥ 5 years; exceptions include the following:

   1. Basal or squamous cell carcinoma of the skin
   2. Carcinoma in situ of the cervix or breast
   3. Incidental histological finding of prostate cancer (Tumour lymphNode Metastasis stage of T1a or T1b)

6. Previous therapy with pomalidomide. 7. Hypersensitivity to thalidomide, lenalidomide, or dexamethasone (this includes ≥ Grade 3 rash during prior thalidomide or lenalidomide therapy).

10. Subjects who are planning for or who are eligible for stem cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-02-28 (Actual); Primary Completion 2017-01-27 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Evaluate efficacy of the combination of pomalidomide and low-dose dexamethasone in subjects with RRMM and impaired renal function | Approximately 2 years
  Overall response rate determined by Myeloma responses determined by modified IMWG criteria

SECONDARY OUTCOMES:
Assessment of renal response according to the criteria defined by Dimopoulos and Ludwig (Dimopoulos, 2009; Dimopoulos, 2010 b,c; Ludwig, 2010). | Approximately 2 years
  Assessment of renal response according to the criteria defined by Ludwig and Dimopoulos
Time to Myeloma response | Approximately 2 years
  Evaluated according to the CTCAE grading
Time to renal response | Approximately 2 years
  Evaluated according to the CTCAE grading
Duration of response | Approximately 2 years
  Evaluated according to the CTCAE grading
Progression-free survival | Approximately 2 years
  Evaluated according to the CTCAE grading
Time to progression | Approximately 2 years
  Evaluated according to the CTCAE grading
Overall Survival | Approximately 2 years
  Evaluated according to the CTCAE grading
Adverse events (AEs) assessment (type, frequency, seriousness, severity, relationship to pomalidomide and/or dexamethasone and outcomes) including second primary malignancy (SPM). | Approximately 2 years
  Pharmacokinetics (PK) of pomalidomide in subjects with RRMM and impaired renal function (moderate to severe renal impairment).

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kueenburg, MD, Study Director — Celgene
Locations (22):
- Austria (3):
  - Krankenhaus der Elisabethinen Linz, I Interne Abteilung, Linz
  - Medizinische Universitat Wien, Vienna
  - Wilhelminenspital der Stadt Wien, Vienna
- France (3):
  - Hopital Dypuytren-CHU de Limoges, Limoges
  - Hopital Saint Louis, Paris
  - CHU de Poitiers, Poitiers
- Germany (2):
  - Medizinische Klinik und Poliklinik V Hamatologie, Onkologie und Rheumatologie, Neuenheimer Feld 410
  - University Hospital Tubingen, Tübingen
- Alexandra Hospital, University of Athens, Athens, Greece
- Italy (4):
  - Azienda Ospedaliero Universitaria Ospedali, Ancona
  - S.C. Oncologia Medica, Lecco
  - Ospedale Maggiore Policlinico Mangiagalli Regina Elena, Milan
  - Arcispedale Santa Maria Nuova, Reggio Emilia
- Netherlands (2):
  - VU University Medical Center VU Medisch Centrum, Amsterdam
  - Daniel den Hoed Kliniek Medical Oncology, Erasmus MC, Rotterdam
- Spain (3):
  - Hospital de La Princesa, Madrid
  - CEIC Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Doctor Peset, Valencia
- United Kingdom (4):
  - Queen Elizabeth Hospital UHB NHS Foundation Trust, Birmingham
  - Ninewells Hospital and Medical School, Dundee
  - Oxford Radcliffe Hospital ICRF Medical Oncology Unit, Headington
  - St Thomas' HospitalGuy's Hospital Dept. of Haematology, London

REFERENCES:
- [Background] Li Y, Wang X, O'Mara E, Dimopoulos MA, Sonneveld P, Weisel KC, Matous J, Siegel DS, Shah JJ, Kueenburg E, Sternas L, Cavanaugh C, Zaki M, Palmisano M, Zhou S. Population pharmacokinetics of pomalidomide in patients with relapsed or refractory multiple myeloma with various degrees of impaired renal function. Clin Pharmacol. 2017 Nov 8;9:133-145. doi: 10.2147/CPAA.S144606. eCollection 2017. PMID 29184451
- [Background] Dimopoulos M, Weisel K, van de Donk NWCJ, Ramasamy K, Gamberi B, Streetly M, Offidani M, Bridoux F, de la Rubia J, Mateos MV, Ardizzoia A, Kueenburg E, Collins S, Di Micco A, Rosettani B, Li Y, Bacon P, Sonneveld P. Pomalidomide Plus Low-Dose Dexamethasone in Patients With Relapsed/Refractory Multiple Myeloma and Renal Impairment: Results From a Phase II Trial. J Clin Oncol. 2018 Jul 10;36(20):2035-2043. doi: 10.1200/JCO.2017.76.1742. Epub 2018 Feb 2. PMID 29394124